CLINICAL TRIAL: NCT02782338
Title: The Effect of Voltaren-ophtha 0.1% (Diclofenac Sodium 0.1%) Eye Drops After Cataract Surgery on INR Levels (International Normalized Ratio) in Patients Taking Warfarin
Brief Title: The Effect of Voltaren-ophtha 0.1% Eye Drops on INR Levels (International Normalized Ratio) in Patients Taking Warfarin
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Lili karmona, Dr., Ophthalmologist, Wolfson Medical Center
Other Study IDs: WolfsonMC
Record Dates: First submitted 2016-05-10; First posted 2016-05-25 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Blood Coagulation Disorders
Keywords: warfarin; Voltaren eye drops; INR
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Voltaren ophtha 0.1% — All study patients will be treated with Voltaren ophtha 0.1% after cataract surgery
  Other Names: voltaren drops

SUMMARY:
A prospective study intended to examine the effect of topical Voltaren-Ophtha 0.1% eye drops after cataract surgery on INR levels (international normalized ratio) in patients taking warfarin.

DETAILED DESCRIPTION:
Objective: To examine the effect of topical Voltaren-Ophtha 0.1% eye drops after cataract surgery on INR levels ( international normalized ratio) in patients taking warfarin.

Methods: A prospective study. The study population will include approximately 100 patients, taking warfarin and that are candidates for cataract surgery. These patients will continue their warfarin therapy as usual and at the same dose, before and after the operation.

INR levels (international normalized ratio) will be checked once a week while taking Voltaren eye drops as is customary after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* people taking warfarin
* candidates for cataract surgery

Exclusion Criteria:

* age <18 years
* pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include approximately 100 patients, taking warfarin and that are candidates for cataract surgery. These patients will continue their warfarin therapy as usual and at the same dose, before and after the operation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
INR levels (international normalized ratio) - change is being assessed | 1 week, 2 weeks, 3 weeks and 4 weeks after taking Voltaren Optha 0.1%
  change is being assessed

IPD SHARING:
Plan to Share IPD: Undecided